CLINICAL TRIAL: NCT02265887
Title: The Pan African Pulmonary Hypertension Cohort Study
Acronym: PAPUCO
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Collaborators: Doula General Hospital, Cameroon (Unknown); Instituto Nacional de Saúde, Mozambique (Other Government); Mayo Clinic (Other); Aminu Kano Teaching Hospital (Other); University of Ibadan (Other); Eduardo Mondlane University (Other); University of Lagos, Nigeria (Other); Khayelitsha District hospital, Cape Town, South Africa (Unknown); Baker Heart Research Institute, Melbourne, Australia (Unknown); Pulmonary Vascular Research Institute, UK (Unknown)
Responsible Party: Principal Investigator, Prof. Karen Sliwa, Professor, University of Cape Town
Other Study IDs: 241/2011
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Africa; Heart Disease; Echocardiography
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Diseases | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: standard of care — No intervention, this a patient registry and is purely an observational study

SUMMARY:
The study will recruit and follow up patients for six months patients newly diagnosed with pulmonary hypertension from twelve centers across four countries; South Africa, Mozambique, Cameroon, Nigeria. The main aim of the study is to describe the aetiology, natural history and management practices of pulmonary hypertension in Africa.

DETAILED DESCRIPTION:
Title: Implementation of the PAPUCO Registry

Background to PAPUCO Registry

The Sub-Saharan Task Force on Pulmonary Hypertension, under the leadership of Dr Ana Olga Mocumbi and Prof. Sliwa, was established in January 2010. The primary aim of this Task Force was to establish a Sub-Saharan African Registry of Pulmonary Hypertension (PHT) and, subsequently, other research and educational awareness projects.

PHT is a devastating, progressive disease, with increasingly debilitating symptoms and, usually, shortened overall life expectancy. The epidemiology of PHT in Sub-Saharan Africa has not yet been determined, but limited reports suggest that the incidence is higher that than reported from developing countries, owing to the pattern of diseases prevalent in the region. Many known factors for PHT are hyperendemic in this part of the world, including Human Immunodeficiency Virus/Acquired Immune Deficiency Syndrome, schistosomiasis, chronic hepatitis B and C and Sickle Cell Disease. On the other hand, a high prevalence of tuberculosis, poorly treated asthma, high levels of pollution in urban areas and exposure to mining, subsequently leads to various forms of pulmonary hypertension and, often, to right heart failure with premature death. Lack of adequate paediatric services to deal with congenital heart disease that leads to pulmonary hypertension, and secondary pulmonary hypertension, is commonly seen, due to the high prevalence of rheumatic heart disease and endomyocardial fibrosis

However, more detailed information is currently not available, thus also leading to poor awareness of those devastating problems, not only in Sub-Saharan Africa, but worldwide. There is, therefore, an urgent need for research into the demographics, natural history and survival of patients with pulmonary hypertension.

Filling these gaps in knowledge is needed to effectively detect, manage and prevent pulmonary hypertension in this region.

The first Sub-Saharan Pulmonary Vascular Hypertension Workshop took place on Friday 23rd and Saturday 24th April 2010, at the Hatter Cardiovascular Research Institute, Chris Barnard Building, Faculty of Health Sciences, University of Cape Town. We had colleagues from South Africa, Africa (Zimbabwe, Mozambique, Nigeria, Kenya, Sudan, Tanzania), United Kingdom (Prof Butrous), Australia (Prof Simon Stewart) and USA (Dr Lori Blauwet) participating in the workshop. The areas of discipline of the participating members ranged from basic scientists, adult and paediatric cardiologists, pulmonologists to cardiothoracic surgeons.

We used the workshop to plan a PHT registry in Africa, under the auspices of the Pulmonary Vascular Research Institute-Sub-Saharan Taskforce.

The main objective of this research is to describe the epidemiology of pulmonary hypertension among patients attending referral units for cardiovascular and pulmonary diseases in African countries. This information will be crucial to the development of effective and resource-sensitive strategies to tackle PHT in Sub-Saharan Africa. The first step in this direction will be to build a registry of patients with PHT, attending a range of hospitals in several countries from this region.

Study Protocol.

Objective: To describe the epidemiology and characteristics of pulmonary hypertension in sub-Saharan Africa

Population:

250 patients with pulmonary hypertension (PHT) who reside in sub-Saharan Africa will be enrolled in the registry.

Each participating center will enroll a minimum of twenty five consecutive patients based on the following eligibility criteria.

Eligibility criteria:

The registry aims to recruit consecutive patients with

1. newly diagnosed PH-based clinical and ECHO criteria,
2. who are able or likely to return for a 6-month follow-up,
3. who are at least 18 years old (except for those in paediatric centres in Mozambique and Nigeria) and
4. who consented in writing to participate in the registry.

Centre eligibility includes

1. availability of ECHO and training in asses- sing right heart function,
2. experience in diagnosing PH according to the WHO classiﬁcation,
3. experience in clinical management of patients with RHF and
4. resources to review patients at 6-month follow-up. Participating centres will be invited to join the registry at African cardiac meetings and conferences.

Recruitment:

Eight centers in 4 countries (Cameroon, Mozambique, Nigeria, South Africa) will recruit patients.

Study Duration:

Recruitment is expected to be complete in 12 to 24 months. Follow-up will continue for a minimum of 6 months after enrollment.

Study Design: This is a prospective observational study.

Study Procedures:

1. Completion of standardized questionnaire to collect epidemiological and clinical data
2. Echocardiographic assessment, including standardized assessment of right ventricular function
3. Collection of peripheral blood for assessment of routine blood investigations and serum biomarkers (in selected centers only, shipment to the Hatter Institute if funding can be secured)
4. Data entry in web-based data system and upload of files as ECG, echocardiography, chest X-ray images. Source documents will be stored at the trial sites.

KEY ROLES

Project Coordinators: Leaders of the Pulmonary Vascular Research Institute Sub-Saharan Africa (PVRI SSA) Task Force [Ana Mocumbi (Mozambique) and Karen Sliwa (Cape Town)] will serve as project coordinators. The Hatter Cardiovascular Research Institute will function as the coordinating centre and will store the serum samples in minus 80 degree freezers.

Principal Investigators: One person from each participating country will be designated to serve as Principal Investigator for that country.

UPDATE 2014 - PUBLICATION:

BMJ Open 2014;4:e005950.doi:10.1136/bmjopen-2014-005950

Rationale and design of the Pan African Pulmonary hypertension Cohort (PAPUCO) study: implementing a contemporary registry on pulmonary hypertension in Africa

Friedrich Thienemann,1,2,3 Anastase Dzudie,3,4 Ana O Mocumbi,5 Lori Blauwet,6 Mahmoud U Sani,7,3 Kamilu M Karaye,7 Okechukwu S Ogah,8,9 Irina Mbanze,10 Amam Mbakwem,11 Patience Udo,12 Kemi Tibazarwa,13 Ahmed S Ibrahim,14 Rosie Burton,15 Albertino Damasceno,10 Simon Stewart,16 Karen Sliwa3,13

Update 2015:

1) Dr Gerald MAARMAN, a member of the PAPUCO group graduated his PhD on animal models of PH at the University of Cape Town (Melatonin as a novel cardioprotective therapy in Pulmonary Hypertension, 2014)

2) Dr Anastase DZUDIE, a Consultant Cardiologist from the Douala General Hospital and investigator of the Cameroon Centre is currently doing his PhD at University of Cape Town. His studies will focus on pulmonary hypertension due to left heart disease. Expected date for submission: August 2015.

3) Dr Friedrich THIENNEMAN presented the Preliminary data analysis after one year of recruitment: the Pan African Pulmonary hypertension Cohort study (PAPUCO) at the Pan African Society of Cardiology Meeting, Dakar, 16th - 19th may 2013.

4) Dr Friedrich THIENNEMAN presented an update of the PAPUCO at the 8th PVRI Annual World Congress; 15-18 January 2015; Guangzhou, China

5) Dr Anastase DZUDIE presented the Clinical profile and outcomes patients with pulmonary hypertension due to left heart disease at the 2nd World Congress on Acute Heart Failure, Seville, 23-26th may 2015.

6) A paper on clinical features and 6 months outcome of group 2 (pulmonary hypertension due to left heat disease) patients in the PAPUCO registry has been submitted in june 2015.

7) An abstract on the "Baseline characteristics and outcome of adult patients included in the PAPUCO registry" : has been accepted for presentation at the forthcoming European Society of Cardiology Congress, London, 29th august-02nd september 2015, UK.

PAPUCO 2 is presently being planned. We envisage recruiting more participants for a long term follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age who meet clinical and echocardiographic criteria for the diagnosis of PHT will be included

Exclusion Criteria:

* Patients who are unable, or unlikely, to return for 6 month follow-up will be excluded

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 250 patients with pulmonary hypertension (PHT) who reside in sub-Saharan Africa will be enrolled in the registry
Sampling Method: Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
mortality | 6 months
  dead or alive status at 6 months post enrolment
To improve performance and functionality | 6 months
  Six minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sliwa-Hahnle, PhD, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Thienemann F, Dzudie A, Mocumbi AO, Blauwet L, Sani MU, Karaye KM, Ogah OS, Mbanze I, Mbakwem A, Udo P, Tibazarwa K, Damasceno A, Keates AK, Stewart S, Sliwa K. The causes, treatment, and outcome of pulmonary hypertension in Africa: Insights from the Pan African Pulmonary Hypertension Cohort (PAPUCO) Registry. Int J Cardiol. 2016 Oct 15;221:205-11. doi: 10.1016/j.ijcard.2016.06.242. Epub 2016 Jun 29. PMID 27404676